CLINICAL TRIAL: NCT04866485
Title: An Open-Label, Phase 1 Clinical Study to Evaluate the Safety, Tolerability, PK/PD and Preliminary Efficacy of HBM4003 in Combination With Anti-PD-1 Monoclonal Antibody in Patients With Advanced NSCLC and Other Solid Tumors
Brief Title: A Study to Evaluate Safety, Tolerability, PK/PD and Preliminary Efficacy of HBM4003 Combined With Anti-PD-1 Antibody
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4003.3
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBM4003+pembrolizumab (Experimental): HBM4003 combined with pembrolizumab in subjects with advanced NSCLC and other solid tumors
  Interventions: Drug: HBM4003 and pembrolizumab

INTERVENTIONS:
Drug: HBM4003 and pembrolizumab — Subjects will be treated with HBM4003 and pembrolizumab on Day 1 during each 21-day cycles.
  Other Names: HBM4003

SUMMARY:
This is an open-label, multi-center phase 1 study. The trial, consisting of Part 1a dose confirmation and Part 1b dose expansion, is designed to evaluate the safety, tolerability, PK/PD and preliminary efficacy of HBM4003 in combination with pembrolizumab in patients with advanced NSCLC and other solid tumors.

DETAILED DESCRIPTION:
subjects will be treated with HBM4003 in combination with pembrolizumab for up to 2 years or until confirmed disease progression, unacceptable tolerability or treatment discontinuation through withdrawal of consent occurs, whichever happens first.

This trial consists of :

* A screening period: 28 days
* A treatment period:

  * Part 1a dose confirmation study
  * Part 1b dose expansion study
* A post-treatment follow-up period, including

  * A safety follow-up period: 28 days after the last dose of study drug;
  * Post-treatment follow-up visit: day 84 after the last dose of study drug;
  * Survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years old at the time of signing the informed consent and ≤ 75 years old at the time of enrollment.
* Patients for Part 1a: patients diagnosed with advanced or recurrent solid tumors.
* Patients for Part 1b: patients diagnosed with metastatic NSCLC and confirmed with negative tumor PD-L1 expression (TPS<1%).
* Patients for Part 1b dose expansion study: have never received systemic therapies as primary therapy for advanced or metastatic diseases.
* Patients must be able to provide fresh tumor tissues or archived tumor tissues.
* Patients whose estimated survival time is more than 3 months.
* Patients with at least one measurable lesion at baseline according to RECIST (version 1.1).
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 1.
* Patients whose organ function must meet the study requirements.
* Males or females with childbearing potential need to use an effective contraceptive method.
* Willing and able to comply with study-specified visits schedule, treatment plan, laboratory examination and other study procedures.

Exclusion Criteria:

* NSCLC patients with EGFR-sensitive mutations or an ALK translocation based on diagnosis results.
* Patients who are simultaneously participating in another clinical study, unless the study is an observational (non-interventional) clinical study or the patient is already in the survival follow-up period of the interventional study.
* Patients with a medical history of severe allergic diseases, a history of severe drug allergies, and are known or suspected allergy to macromolecular protein preparations or HBM4003 or pembrolizumab excipients.
* Previous and concomitant drugs or treatments to be excluded like CTLA4, PD-1,PD-L1.
* Insufficient completely recovery from previous treatments.
* Diseases that may affect the efficacy and safety of the investigational product.
* A history of other malignant diseases within 5 years before the first dose.
* Active brain metastasis or leptomeningeal metastasis during screening or previous with imaging evidence (based on CT or MRI assessment).
* Patients who have received palliative radiotherapy for non-central nervous system lesions within 2 weeks before the first dose.
* Patients who have received more than 30 Gy of lung radiation therapy within 6 months before the first dose.
* A history of interstitial lung disease or non-infectious pneumonia.
* Patients with pleural effusion, pericardial effusion, or ascites.
* Patients that may have other conditions that affect the efficacy or safety evaluation of this study (such as mental disorder, alcoholism, drug abuse, etc.) .
* Women who are pregnant or breastfeeding, or who plan to become pregnant during the study period and within 3 months after the last dose of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-06-14 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Part 1a: Number of subjects with DLT in each dose group within 1 cycles (21 days) after the first drug administration | approximate 21 days
  DLT observation period was defined as one treatment cycles with a total of 21 days
Part 1b: ORR | maximum 2 years
  Proportion of subjects with complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Part 1a: ORR | maximum 2 years
  including proportions of subjects with complete response (CR) and partial response (PR)
Part 1a: Disease Control Rate, DCR | maximum 2 years
  including proportion of subjects with complete response (CR) and partial response (PR) and stable disease (SD)
Part 1a: Duration of Response, DOR | maximum 2 years
  Calculate the duration from the first confirmed CR or PR to the date of disease progression or death (for any reason)
Part 1a: Duration of Disease Control, DDC | maximum 2 years
  For subjects with Cr, PR or SD, the duration from the time of initial administration to the date of disease progression or death (for any reason) was calculated
Cmax | maximum 2 years
  Peak Plasma Concentration
Tmax | maximum 2 years
  Time to reach maximum serum concentration
AUC0-last | maximum 2 years
  Area under the plasma concentration versus time curve from time zero to last
AUC0-tau | maximum 2 years
  Area under the serum concentration versus time curve from time zero to the dosing interval tau
UC0-inf | maximum 2 years
  Area under the serum concentration versus time curve from time zero to infinity
Vss | maximum 2 years
  Volume of distribution at steady state
CL | maximum 2 years
  Clearance
t1/2 | maximum 2 years
  Terminal half-life
Part 1a: Immunogenicity of HBM4003 and pembrolizumab | maximum 2 years
  including the occurrence of positive anti-drug antibodies (ADA). The occurrence of neutralizing antibodies for subjects with positive ADA
Part 1b: Number of subjects experiencing at least one treatment-related AE | maximum 2 years
  Evaluate safety
Part 1b: DCR | maximum 2 years
  including proportion of subjects with CR, PR and SD
Part 1b: DOR | maximum 2 years
  calculate the duration from the first confirmed CR or PR to the date of disease progression or (for any reason) death.
Part 1b: DDC | maximum 2 years
  for subjects with CR, PR or SD, calculate the duration from the time of initial medication to the day of disease progression or (for any reason) death
Part 1b: Overall survival (OS) | maximum 2 years
  the length of time from the start of treatment to the death of the subject (for any reason)
Part 1b: Progression-free survival (PFS) | maximum 2 years
  the length of time from the beginning of treatment to the beginning of disease progression or death (for any reason)
Part 1b: Immunogenicity of HBM4003 and pembrolizumab | maximum 2 years
  including the occurrence of positive anti-drug antibodies (ADA). The occurrence of neutralizing antibodies for subjects with positive ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Shun LU, Doctor, Principal Investigator — Shanghai Chest Hospital